CLINICAL TRIAL: NCT04951128
Title: The Effect of Local Tranexamic Acid on Post-operative Edema and Ecchymosis in Eyelid Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Consultants in Ophthalmic and Facial Plastics Surgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Tranexamic Acid
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Edema; Ecchymosis; Eyelid
Keywords: Tranexamic acid; Post-operative ecchymosis; Post-operative edema
MeSH Terms: conditions — Edema; Ecchymosis | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants in this study will undergo bilateral upper/lower eyelid surgery. The treatment side with tranexamic acid will be randomized for each patient using a random coin flip generator (head for the right side and tail for left side). The surgeons, participants, and photo reviewers will be blinded to the treatment side.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid arm (Experimental): Eyelid(s) that received tranexamic acid in the local anesthetic
  Interventions: Drug: Tranexamic acid injection
- Control (Active Comparator): Eyelid(s) that receive local anesthetic without tranexamic acid
  Interventions: Other: Local anesthetic control

INTERVENTIONS:
Drug: Tranexamic acid injection — Tranexamic acid (100 mg/mL concentration; 0.5 mL) will be added to local anesthetic mixture of 2% lidocaine with epinephrine (2.25 mL) and 0.5% bupivacaine with epinephrine (2.25mL).
  Arms: Tranexamic acid arm
Other: Local anesthetic control — Local anesthetic mixture without tranexamic acid consisting of 2% lidocaine with epinephrine (2.5 mL) and 0.5% bupivacaine with epinephrine (2.5 mL).
  Arms: Control

SUMMARY:
Tranexamic acid (TXA) is a synthetic inhibitor of plasminogen lysine receptor that has used to reduce intra-operative bleeding in a number of clinical scenarios. Anecdotally, TXA has used by plastic surgeons to reduce post-operative bruising. To date, there is limited data to valid the benefits and to evaluate the side effects of TXA. The objective of this study is to evaluate the effect of local TXA on edema and ecchymosis in eyelid surgery.

DETAILED DESCRIPTION:
Tranexamic acid (TXA) is a synthetic reversible competitive inhibitor to plasminogen lysine receptor, which prevents plasmin formation and stabilizes the fibrin matrix, thus reduce bleeding. Recent studies have demonstrated the antifibrinolytic benefits of TXA in a number of clinical scenarios, including heavy menstrual bleeding, traumatic hemorrhage, elective cesarean section, total knee arthroplasty, coronary artery surgery, spinal deformity surgery, orthognathic surgery, transurethral prostate resection, aneurysmal subarachnoid hemorrhage, epistaxis, and hemoptysis.

Anecdotally, TXA has been used by plastic surgeons to reduce postoperative bruising. However, there is a paucity of clinical data on TXA use in plastic surgery, and the results are inconsistent. In a prospective randomized controlled trial evaluating local TXA in upper blepharoplasty, Sagiv et al reported no intraoperative blood loss, surgeon's assessment of hemostasis, and periocular ecchymosis size on postoperative day 1. Butz and Geldner reviewed their experience placing TXA-soaked pledgets in 57 patients who underwent face lift18. They identified only 1 patient who had post-operative hematoma and they reported no systemic complications from TXA use. In a randomized control trial evaluating topical TXA in reduction mammoplasty, Ausen et al reported 39% reduction of postoperative fluid drainage on the treatment side. In a study evaluating oral TXA and cortisone effect in rhinoplasty, Sakalliogu et al reported significant reduction of intraoperative bleeding and postoperative ecchymosis/edema in patients who underwent rhinoplasty. Further study is warranted to evaluate the use to TXA in plastic surgery. The objective of this study is to evaluate the effect of local TXA on edema and ecchymosis in eyelid surgery.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* Undergo bilateral upper/lower eyelid blepharoplasty, bilateral upper eyelid ptosis repair, or a combination of the above procedures
* Additional concurrent forehead/brow or upper/lower eyelids surgeries may be included if bilateral

Exclusion Criteria:

* Prior eyelid surgery
* Anticoagulant or antiplatelet use, including aspirin, within 7 days prior to surgery
* Patient who is currently pregnant or breast feeding
* Patient with color vision deficiency
* TXA allergy
* History of bleeding disorder
* History of clotting disorder
* History of seizure
* Have active nausea/vomiting/gastrointestinal symptoms
* Have active intracranial bleeding
* Have active periocular ecchymosis or edema prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative edema/ecchymosis | 1st post op visit: post-op day 1 to 3
  Post-operative edema/ecchymosis will be graded by Winkler-Black Bruising Scale (0= no bruising, 1= mild bruising, 2=moderate bruising, 3=severe bruising)
Post-operative edema/ecchymosis | 2nd post op visit: post-op day 7 to 10
  Post-operative edema/ecchymosis will be graded by Winkler-Black Bruising Scale (0= no bruising, 1= mild bruising, 2=moderate bruising, 3=severe bruising)

SECONDARY OUTCOMES:
Post-operative complications | 1st post op visit: post-op day 1 to 3
  Potential complications: allergic reaction, persistent bleeding, thromboembolic event, wound dehiscence, wound infection, or tissue necrosis
Post-operative complications | 2nd post op visit: post-op day 7 to 10
  Potential complications: allergic reaction, persistent bleeding, thromboembolic event, wound dehiscence, wound infection, or tissue necrosis

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Consultants in Ophthalmic and Facial Plastic Surgery, Southfield, Michigan
  - Montefiore Medical Center, The Bronx, New York
  - Houston Methodist, Houston, Texas
  - University of Texas - Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rohrich RJ, Cho MJ. The Role of Tranexamic Acid in Plastic Surgery: Review and Technical Considerations. Plast Reconstr Surg. 2018 Feb;141(2):507-515. doi: 10.1097/PRS.0000000000003926. PMID 28938364
- [Background] Lukes AS, Moore KA, Muse KN, Gersten JK, Hecht BR, Edlund M, Richter HE, Eder SE, Attia GR, Patrick DL, Rubin A, Shangold GA. Tranexamic acid treatment for heavy menstrual bleeding: a randomized controlled trial. Obstet Gynecol. 2010 Oct;116(4):865-875. doi: 10.1097/AOG.0b013e3181f20177. PMID 20859150
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] CRASH-2 collaborators; Roberts I, Shakur H, Afolabi A, Brohi K, Coats T, Dewan Y, Gando S, Guyatt G, Hunt BJ, Morales C, Perel P, Prieto-Merino D, Woolley T. The importance of early treatment with tranexamic acid in bleeding trauma patients: an exploratory analysis of the CRASH-2 randomised controlled trial. Lancet. 2011 Mar 26;377(9771):1096-101, 1101.e1-2. doi: 10.1016/S0140-6736(11)60278-X. PMID 21439633
- [Background] Morrison JJ, Dubose JJ, Rasmussen TE, Midwinter MJ. Military Application of Tranexamic Acid in Trauma Emergency Resuscitation (MATTERs) Study. Arch Surg. 2012 Feb;147(2):113-9. doi: 10.1001/archsurg.2011.287. Epub 2011 Oct 17. PMID 22006852
- [Background] Gungorduk K, Yildirim G, Asicioglu O, Gungorduk OC, Sudolmus S, Ark C. Efficacy of intravenous tranexamic acid in reducing blood loss after elective cesarean section: a prospective, randomized, double-blind, placebo-controlled study. Am J Perinatol. 2011 Mar;28(3):233-40. doi: 10.1055/s-0030-1268238. Epub 2010 Oct 26. PMID 20979013
- [Background] Alvarez JC, Santiveri FX, Ramos I, Vela E, Puig L, Escolano F. Tranexamic acid reduces blood transfusion in total knee arthroplasty even when a blood conservation program is applied. Transfusion. 2008 Mar;48(3):519-25. doi: 10.1111/j.1537-2995.2007.01564.x. Epub 2007 Dec 7. PMID 18067499
- [Background] Gomez-Barrena E, Ortega-Andreu M, Padilla-Eguiluz NG, Perez-Chrzanowska H, Figueredo-Zalve R. Topical intra-articular compared with intravenous tranexamic acid to reduce blood loss in primary total knee replacement: a double-blind, randomized, controlled, noninferiority clinical trial. J Bone Joint Surg Am. 2014 Dec 3;96(23):1937-44. doi: 10.2106/JBJS.N.00060. PMID 25471907
- [Background] Myles PS, Smith JA, Forbes A, Silbert B, Jayarajah M, Painter T, Cooper DJ, Marasco S, McNeil J, Bussieres JS, McGuinness S, Byrne K, Chan MT, Landoni G, Wallace S; ATACAS Investigators of the ANZCA Clinical Trials Network. Tranexamic Acid in Patients Undergoing Coronary-Artery Surgery. N Engl J Med. 2017 Jan 12;376(2):136-148. doi: 10.1056/NEJMoa1606424. Epub 2016 Oct 23. PMID 27774838
- [Background] Choi HY, Hyun SJ, Kim KJ, Jahng TA, Kim HJ. Effectiveness and Safety of Tranexamic Acid in Spinal Deformity Surgery. J Korean Neurosurg Soc. 2017 Jan 1;60(1):75-81. doi: 10.3340/jkns.2016.0505.004. Epub 2016 Dec 29. PMID 28061495
- [Background] Choi WS, Irwin MG, Samman N. The effect of tranexamic acid on blood loss during orthognathic surgery: a randomized controlled trial. J Oral Maxillofac Surg. 2009 Jan;67(1):125-33. doi: 10.1016/j.joms.2008.08.015. PMID 19070758
- [Background] Kumsar S, Dirim A, Toksoz S, Saglam HS, Adsan O. Tranexamic acid decreases blood loss during transurethral resection of the prostate (TUR -P). Cent European J Urol. 2011;64(3):156-8. doi: 10.5173/ceju.2011.03.art13. Epub 2011 Sep 6. PMID 24578884
- [Background] Rannikko A, Petas A, Taari K. Tranexamic acid in control of primary hemorrhage during transurethral prostatectomy. Urology. 2004 Nov;64(5):955-8. doi: 10.1016/j.urology.2004.07.008. PMID 15533485
- [Background] Hillman J, Fridriksson S, Nilsson O, Yu Z, Saveland H, Jakobsson KE. Immediate administration of tranexamic acid and reduced incidence of early rebleeding after aneurysmal subarachnoid hemorrhage: a prospective randomized study. J Neurosurg. 2002 Oct;97(4):771-8. doi: 10.3171/jns.2002.97.4.0771. PMID 12405362
- [Background] Zahed R, Mousavi Jazayeri MH, Naderi A, Naderpour Z, Saeedi M. Topical Tranexamic Acid Compared With Anterior Nasal Packing for Treatment of Epistaxis in Patients Taking Antiplatelet Drugs: Randomized Controlled Trial. Acad Emerg Med. 2018 Mar;25(3):261-266. doi: 10.1111/acem.13345. Epub 2017 Dec 9. PMID 29125679
- [Background] Wand O, Guber E, Guber A, Epstein Shochet G, Israeli-Shani L, Shitrit D. Inhaled Tranexamic Acid for Hemoptysis Treatment: A Randomized Controlled Trial. Chest. 2018 Dec;154(6):1379-1384. doi: 10.1016/j.chest.2018.09.026. Epub 2018 Oct 12. PMID 30321510
- [Background] Sagiv O, Rosenfeld E, Kalderon E, Barazani TB, Zloto O, Martinowitz U, Ben Simon GJ, Zilinsky I. Subcutaneous tranexamic acid in upper eyelid blepharoplasty: a prospective randomized pilot study. Can J Ophthalmol. 2018 Dec;53(6):600-604. doi: 10.1016/j.jcjo.2018.01.006. Epub 2018 Mar 27. PMID 30502984
- [Background] Butz DR, Geldner PD. The Use of Tranexamic Acid in Rhytidectomy Patients. Plast Reconstr Surg Glob Open. 2016 May 25;4(5):e716. doi: 10.1097/GOX.0000000000000745. eCollection 2016 May. No abstract available. PMID 27579240
- [Background] Ausen K, Fossmark R, Spigset O, Pleym H. Randomized clinical trial of topical tranexamic acid after reduction mammoplasty. Br J Surg. 2015 Oct;102(11):1348-53. doi: 10.1002/bjs.9878. PMID 26349843
- [Background] Sakallioglu O, Polat C, Soylu E, Duzer S, Orhan I, Akyigit A. The efficacy of tranexamic acid and corticosteroid on edema and ecchymosis in septorhinoplasty. Ann Plast Surg. 2015 Apr;74(4):392-6. doi: 10.1097/SAP.0b013e3182a1e527. PMID 24149401
- [Background] Wellington K, Wagstaff AJ. Tranexamic acid: a review of its use in the management of menorrhagia. Drugs. 2003;63(13):1417-33. doi: 10.2165/00003495-200363130-00008. PMID 12825966
- [Background] Berntorp E, Follrud C, Lethagen S. No increased risk of venous thrombosis in women taking tranexamic acid. Thromb Haemost. 2001 Aug;86(2):714-5. No abstract available. PMID 11522029
- [Background] Lindoff C, Rybo G, Astedt B. Treatment with tranexamic acid during pregnancy, and the risk of thrombo-embolic complications. Thromb Haemost. 1993 Aug 2;70(2):238-40. PMID 8236125
- [Background] Tavakoli N, Mokhtare M, Agah S, Azizi A, Masoodi M, Amiri H, Sheikhvatan M, Syedsalehi B, Behnam B, Arabahmadi M, Mehrazi M. Comparison of the efficacy of intravenous tranexamic acid with and without topical administration versus placebo in urgent endoscopy rate for acute gastrointestinal bleeding: A double-blind randomized controlled trial. United European Gastroenterol J. 2018 Feb;6(1):46-54. doi: 10.1177/2050640617714940. Epub 2017 Jun 20. PMID 29435313